CLINICAL TRIAL: NCT03265756
Title: Multimometer - Vital Signs Device for Diagnosis of Pneumonia
Status: Completed | Type: Observational
Sponsor: University of Alberta (Other)
Collaborators: Grand Challenges Canada (Other)
Responsible Party: Principal Investigator, Israel Amirav, MD, University of Alberta
Other Study IDs: Pro00072555
Record Dates: First submitted 2017-08-26; First posted 2017-08-29 (Actual); Last update posted 2018-11-21 (Actual); Status verified 2018-11

CONDITIONS: Pneumonia
MeSH Terms: conditions — Pneumonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy children: 250 3D facial images of healthy children under 5yrs of age in the Democratic Republic of Congo (DRC).
- Suspected Pneumonia: 50 young children (under 5 yrs) in hospital/clinics in Butembo DRC with suspected pneumonia
  Interventions: Device: Multimometer

INTERVENTIONS:
Device: Multimometer — A device for measuring respiration rate, temperature, heart rate and the degree of blood oxygenation of children
  Groups: Suspected Pneumonia

SUMMARY:
Pneumonia is a major cause of illness in young children. The investigators are developing and testing a new thermometer like device called Multimometer, to measure the respiration rate (RR), temperature, heart rate (HR) and the degree of blood oxygenation (SpO2) of children who may suffer from pneumonia. These are called vital signs and their measurements greatly help to diagnose pneumonia.

In the first part of the study, and in order to optimize and better align the size of the device with the face, the investigators will measure the average size and dimensions of young children's face. In the second part of the study, the investigators will compare the vital signs measurements with measurements obtained by other commonly used devices in ill children who are suspected to suffer from pneumonia.

DETAILED DESCRIPTION:
A. Improve the universality of the mouth-interface using facial anthropometry techniques.

For this first part of the study, the investigators will use a portable 3D camera (as previously used by our group) to acquire 250 3D facial images of healthy children under 5yrs of age in the DRC. While in hospital/clinic, the investigators will use a three-dimension (3D) special camera to obtain an image of the child's face. The child can sit on the lap of the parent and we will take the image. The image acquisition takes less than 30 seconds. There are no specific requirements from the child, and the image can be taken if the child is asleep or awake, cry or settled. No medical or identifying information will be collected.

All the computerized images will be cluster analyzed (using previously established methodologies from the Technion, Israel) and three 3D average faces of all small, medium and large faces will be constructed. The investigators will use these "faces" to design better Multimometers with improved mouth-interface for this population.

B. Integrate into the current device a reflexive pulse oximeter sensor which will allow measurements of oxygen saturation and heart rate.

For the addition of HR and SpO2 measurements, the investigators will integrate a reflective pulse oximetry chip into the probe. Together with the manufacturer (RespiDx Inc., Israel) the investigators will design and manufacture optimal prototype devices suitable for performing clinical trials on this population.

C. Compare vital signs measurements by Multimometer® to simultaneous vital signs measurement using conventional devices.

For this part of the study, repeated (x5 times) measurements of the 4 vital signs in 50 young children (under 5 yrs) in hospital/clinics in Butembo DRC with suspected pneumonia, will be recorded using the Multimometer. These signs will also be measured at the same time, by conventional methods (regular thermometers for temperature, observed respiratory rate using recorded chest movements and end-tidal carbon dioxide (CO2) for respiratory rate, standard pulse oximeters for oxygen saturation and heart rate). All these measurements take less than 5 minutes. The investigators will repeat these sets approximately 5 times during the same day in the hospital or during a clinic visit. The vital signs will be compared between the two methods using Pearson's correlation coefficient and using Bland-Altman plots for agreement.

ELIGIBILITY:
Inclusion Criteria:

For the first part of the study (3D facial images):

• Healthy children under 5y of age

For the second phase of the study (Comparison of vital signs):

• Children under 5y of age with suspected pneumonia

Exclusion Criteria:

• Children older than 5y of age

Max Age: 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children under 5y of age
Sampling Method: Non-Probability Sample
Enrollment: 350 (Actual)
Dates: Start 2017-06-20 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
Vital Signs Comparison | 2018
  Measurements of respiration rate, temperature, heart rate and the degree of blood oxygenation of children

SECONDARY OUTCOMES:
3D facial images | 2017-2018
  Measurements of facial dimensions and contour

CONTACTS AND LOCATIONS:
Overall Officials: Israel Amirav, Principal Investigator — University of Alberta
Locations (2):
- University of Alberta, Edmonton, Alberta, Canada
- AHFIA (Association for Health Innovation in Africa), Butembo, North Kivu, Democratic Republic of the Congo

IPD SHARING:
Plan to Share IPD: Undecided